CLINICAL TRIAL: NCT06019780
Title: Effects of Blood Flow Restriction Training in Patients With Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU Hina Yasmeen
Record Dates: First submitted 2023-08-26; First posted 2023-08-31 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive capsulitis; Blood flow restriction training; Range of motion
MeSH Terms: conditions — Bursitis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental interventional group A (Blood flow restriction training) (Experimental): Following exercise will be performed
  1. Side lying external rotation
  2. Prone horizontal abduction
  3. Standing scaption with pneumatic cuff for blood flow restriction
  Interventions: Other: blood flow restriction trainin
- Control group B (Active Comparator): Following exercise will be performed
  1. Side lying external rotation
  2. Prone horizontal abduction
  3. Standing scaption without blood flow restriction
  Interventions: Other: exercise

INTERVENTIONS:
Other: blood flow restriction trainin — Following exercise will be performed
  1. Side lying external rotation
  2. Prone horizontal abduction
  3. Standing scaption İndividual in the group will be having two session per week, 16 session of exercise training for 8 weeks.50% of arterial occlusion pressure (60 to 80 mmHg) will be applied for total duration of 15mins. Occlusion pressure will be calculated according to formula for each patient [Pressure=0.4x(systolic BP)+2.7x(shoulder circumference)+62].4 sets with one set of 30 repetition and three sets of 15 repetition. After each set subject will have 30 seconds of rest with cuff inflated.
  Arms: Experimental interventional group A (Blood flow restriction training)
Other: exercise — Following exercises will be performed without application of pneumatic cuff
  1. Side lying external rotation
  2. Prone horizontal abduction
  3. Standing scaption Conventional treatment will include: Hot pack 5 mins Maitland grade 3 and 4 mobilization: inferior glide (10reps x3sets), posterior glide (10reps x 3sets), anterior glide (10 reps x 3sets) Home plan: wand exercise, pendulum exercise, wall walking exercise (10reps x 2sets each)
  Arms: Control group B

SUMMARY:
The aim of this research is to determine the effect of blood flow restriction training on shoulder pain, range of motion, muscle strength and shoulder. Randomized controlled trials will be done at Lady Reading Hospital Peshawar and Shahab Orthopedic General Hospital. The sample size is 36. The subjects will be divided in two groups, 18 subjects in BFR group and 18 in no BFR group. Study duration is 6 months. Sampling technique applied was non probability connivance sampling technique. Tools used in the study are SPADI shoulder score, NPRS, hand held dynamometer, sphygmomanometer and goniometer.

DETAILED DESCRIPTION:
Frozen shoulder is painful shoulder condition associated with stiffness and shoulder disability. It is associated with reduction in forward elevation and marked external rotation. Frozen shoulder is common condition effecting population between ages 30 to 60 years. Prevalence is more common in women than on men There are four stages of adhesive capsulitis, stage1, stage 2 (freezing stage), stage 3 (frozen stage) and stage 4 (thawing stage). Patient have sharp pain at end range of motion, sleep disturbances and early loss of external rotation. When compared to asymptomatic subjects, patients with adhesive capsulitis have higher upper trapezius to lower trapezius EMG ratios during arm elevation, indicating a muscular imbalance. The scapula eventually migrates upward before 60 degrees of abduction in individuals with adhesive capsulitis, resulting in the recognizable "shrug sign" during shoulder elevation.

Blood flow is restricted in a controlled form of vascular occlusion using external tourniquet. A recent study demonstrated that augmentation of low load resistance with blood flow restriction (L-L BFR) to contractile tissue can produce hypertrophy and strength gains, using loads as low as 30% 1RM. BFR exercise may stimulate skeletal muscle growth and strength gains through a number of different methods. These could include an increase in hormone levels, an increase in the motor pathway or other intracellular signaling pathways for muscle protein synthesis, an increase in satellite cell activity biomarkers, and apparent patterns in fibre type recruitment.

The purpose of this study is to provide the effects of blood flow restriction training on shoulder discomfort, range of motion, muscle strength and disability in patients with adhesive capsulitis. Due to pain and decrease range of motion individual with adhesive capsulitis experience muscle weakness in shoulder joint. Blood flow restriction training has positive effect on improvement of muscle strength and range of motion in shoulder region. Blood flow restriction training has also positive effect on bone healing and bone density. Therefore the study is aimed to improve the muscles strength and capsule inflammation in individual with adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Frozen shoulder (stage 2 and 3 of Kisner and Colby's classification system)
* Male and female
* Patients whose age lies between 40 and 60
* Ranges restriction in forward flexion (scaption) less than 100 degree and reduction of external and internal rotation to less than 50% of the normal

Exclusion Criteria:

* • History of Cardiovascular diseases

  * DVT patients
  * Hypertensive patients
  * Patients having neurological disease
  * Fracture of humerus

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
shoulder apin | baseline to 4th to 8 weeks
  the shoulder pain will be measured by NPRS, it has 11 points with 0 no pain and 10 extreme pain.
Shoulder flexors strength | baseline to 8 weeks
  this will be measured by the dynamometer by placing the dynamometer over the muscles and the individual will apply flexion force against isometric resistance.
Shoulder extensors strength | baseline to 8 weeks
  this will be measured by the dynamometer by placing the dynamometer over the muscles and the individual will apply extension force against isometric resistance.
Shoulder abductors strength | baseline to 8 weeks
  this will be measured by the dynamometer by placing the dynamometer over the muscles and the individual will apply abduction force against isometric resistance.
Shoulder rotation strength | baseline to 8 weeks
  this will be measured by the dynamometer by placing the dynamometer over the muscles and the individual will apply rotation force against isometric resistance.
Shoulder disability (SPADI) | baseline to 8 weeks
  measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.

SECONDARY OUTCOMES:
shoulder flexion | baseline to 8 weeks
  measures the shoulder flexion range of motion through goniometry
Shoulder extension | baseline to 8 weeks
  measures the shoulder extension range of motion through goniometry
shoulder abduction | baseline to 8 weeks
  measures the shoulder abduction range of motion through goniometry
shoulder adduction | baseline to 8 weeks
  measures the shoulder adduction range of motion through goniometry
shoulder internal rotation | baseline to 8 weeks
  measures the shoulder internal rotation range of motion through goniometry
shoulder external rotation | baseline to 8 weeks
  measures the shoulder external rotation range of motion through goniometry

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Shahab orthopedic general hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No